CLINICAL TRIAL: NCT02873351
Title: Pilot Study of L-DOPA Safety and Tolerability in Patients With AMD, and Proof of Concept That L-DOPA Improves Surrogate Biomarkers in Patients With Moderate to Advanced AMD
Brief Title: A Safety and Efficacy Study of Carbidopa-levodopa in Patients With Macular Degeneration
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decided to do studies in patients with AMD
Sponsor: Snyder, Robert W., M.D., Ph.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000
Record Dates: First submitted 2016-07-26; First posted 2016-08-19 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2017-05

CONDITIONS: Age-related Macular Degeneration
Keywords: L-DOPA; GPR143; PEDF; VEGF
MeSH Terms: conditions — Macular Degeneration | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- carbidopa-levodopa 25-100 mg (Experimental): Treatment with carbidopa-levodopa 25-100 mg tablets dosed once daily at bedtime for 45 +/- 5 days followed by carbidopa-levodopa 25-100 mg tablets dosed 3 times daily for 45 +/- 5 days.
  Interventions: Drug: carbidopa-levodopa 25-100 mg
- Placebo for carbidopa-levodopa 25-100 mg (Placebo Comparator): Treatment with placebo for carbidopa-levodopa 25-100 mg in identical tablets dosed once daily at bedtime for 45 +/- 5 days followed by placebo for carbidopa-levodopa 25-100 mg tablets dosed 3 times daily for 45 +/- 5 days.
  Interventions: Drug: placebo for carbidopa-levodopa 25-100 mg

INTERVENTIONS:
Drug: carbidopa-levodopa 25-100 mg — included in arm description
  Arms: carbidopa-levodopa 25-100 mg
Drug: placebo for carbidopa-levodopa 25-100 mg — included in arm description
  Arms: Placebo for carbidopa-levodopa 25-100 mg

SUMMARY:
From 3 large patient databases, patients diagnosed with AMD who have never taken levodopa(L-DOPA) containing medications have a mean age of diagnosis at 71 years. Patients who have been treated with L-DOPA containing medications have a mean age of diagnosis of AMD at 79 years.

L-DOPA binds to GPR143 in the retinal pigment epithelium, and releases PEDF, which protects the retina and downregulates VEGF, which is the cause of neovascularization.

The Investigators will evaluate the safety and tolerability of carbidopa-levodopa in patients with AMD, and measure the effects on surrogate functional biomarkers of AMD.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the most common cause of blindness, in individuals over the age of 50, in the developed world(1,2). AMD becomes more common as people age, and is more common in lightly pigmented individuals(3). AMD appears more common in patients with Parkinson's Disease, than in those without(4). The AREDS nutritional supplements are effective in slowing the progress of intermediate AMD(5). Most AMD is "dry AMD", which progresses relatively slowly and may impair vision, but usually does not lead to legal blindness. There are two forms of AMD, "wet AMD" and geographic atrophy (GA), that can cause more profound vision loss. In aggregate they occur in about 25% patients with AMD(5). Wet AMD is due to new growth of abnormal blood vessels under the retina. The new blood vessels are believed to be due to an excessive release of vascular endothelial growth factor (VEGF) by the retinal pigment epithelium(RPE) cells(6). Wet AMD is now effectively treated with intraocular injections of VEGF inhibitors(2). Geographic Atrophy, the other form of advanced AMD, represents focal death of the RPE cells and overlying neurosensory retina. There is no current treatment for GA. It is suspected that GA is due in part to a localized inflammatory response, damage to RPE cells and loss of RPE cell function(7). It may also be speculated that stimulation of RPE cells to release a potent neurotrophic factor, pigment epithelium derived factor (PEDF) may slow progression of GA.

In 2008, Dr. Brian McKay identified a receptor, G protein coupled receptor #143(GPR143), on the surface of RPE cells and discovered that L-DOPA was the natural ligand or stimulator of GPR143(8). Dr McKay showed that treatment of RPE cells with exogenous L-DOPA resulted in the release of additional PEDF. In subsequent work Dr McKay's group also showed that L-DOPA stimulation of PEDF in RPE cells was also associated with a decrease in VEGF(9). Thus, Dr McKay hypothesized that exogenous L-DOPA may prevent the onset of AMD or progression to wet AMD.

In 2015, Dr McKay and his associates published a paper that showed that patients, who had been treated with L-DOPA, had a delay in the onset of AMD by 8 years, compared to patients who had not been treated with L-DOPA(10). In addition, those who had AMD and went on to develop wet AMD, did so 5 years later than those with no history of L-DOPA treatment(10). L-DOPA is an intermediate in the pigmentation pathway. Dr McKay and his associates suggested that the reason darkly pigmented races do not get AMD nearly as frequently as lighter pigmented races, is that they produce more pigment, and thus more L-DOPA to stimulate GPR143 on RPE cells. According to this hypothesis, the stimulated RPE cells release PEDF and decrease VEGF, which together are responsible for the protective effect.

Since there are no established animal models for AMD, and L-DOPA has a good safety profile in healthy volunteers and patients with Parkinson's disease(11), the Investigators propose a prospective experiment to determine the safety and tolerability of L-DOPA, in a population of patients with AMD. The participants will be made aware of potential side effects of L-DOPA, which are listed in the Informed Consent, during the consent process. Adverse events will be elicited by questioning the participants at each visit. The participants will also be advised to call the site, if they have any medical problem between visits.

The Investigators will also use this safety study to examine whether L-DOPA has a positive effect on surrogate biomarkers of AMD. The surrogate markers to be evaluated are dark adaptation(12,13), best corrected visual acuity (BCVA), low luminance visual acuity(LLVA)(14), and the size and numbers of drusen(15) and reticular pseudodrusen(16). A previous trial, with retinol in 104 patients, significantly improved dark adaptation in 30 days.(17) Therefore, the Investigators expect to see improvement with L-DOPA in a relatively short time. This study will also help the Investigators prepare for a Phase 3 study of L-DOPA in AMD.

Pharmacology of L-DOPA and carbidopa

L-DOPA is formed by 3-hydroxylation of tyrosine by tyrosine-3-monooxygenase (tyrosinase).(18) The primary metabolic pathway of L-DOPA is decarboxylation by amino acid decarboxylase to dopamine, which is responsible for most, but not all, of its pharmacologic effects and toxicity. When carbidopa is administered with L-DOPA, systemic levels of L-DOPA double and central nervous system (CNS) L-DOPA increases from about 1% of the administered dose to about 4%. Levodopa freely passes from the systemic circulation into the retina and brain, but dopamine and carbidopa do not. Adverse events are markedly decreased when carbidopa is administered with L-DOPA, because systemic levels of the toxic metabolite of L-DOPA, dopamine, are markedly reduced. In most patients, 25 mg of carbidopa is sufficient to control side effects of 100 mg of L-DOPA, primarily nausea(18), by 90%. However, some patients require additional supplemental carbidopa. Carbidopa has very limited side effects when given alone(18). Therefore, the Investigators plan to use 35 mg of carbidopa with each 100 mg of levodopa, in order to control adverse events in almost all participants.

L-DOPA is the natural ligand for GPR143 in the RPE cells(8). The Investigators' intent is to increase the L-DOPA available to RPE surface receptors (GPR 143) while minimizing peripheral toxicity. This concept is unique, because all other uses of L-DOPA rely on CNS conversion of L-DOPA to dopamine, in order to produce the desired effect(19).

Treatments:

1. Carbidopa-levodopa 35-100 mg dosed hs for 45 days, followed by carbidopa-levodopa 35-100 mg dosed in the morning, with supper and hs for 45 days. The second dosing period is the equivalent of a moderate dose of carbidopa-levodopa in patients with Parkinson's disease (maximum daily dose 200-800 mg).
2. Placebo dosed hs for 45 days, followed by placebo dosed in the morning, with supper and hs for 45 days.

Placebo and active medication will be dosed as capsules, identical in appearance.

Number of participants: Not yet recruiting, stratified by non-study eye being normal, dry AMD or wet AMD and randomized using a table of random numbers. Estimated screen failure rate is 50%. The sample size is based on a successful study treating patients with impaired dark adaptation with retinol, which showed significant improvement in 30 days with 52 patients per study arm.

Duration: 87-114 days (80-100 days of treatment). Visits 1 (screening) and 2(randomization) can be scheduled within 1 week. The first visit after Randomization, Visit 3, will occur 40-50 days after Visit 2. Visit 4 (end of study) will occur 40-50 days after Visit 3. This schedule allows a 10 day window for study visits, for logistic reasons and patient convenience.

Overall trial duration for enrollment and treatment, screening 5 patients per week, will be approximately 10 months.

Primary Endpoint: A statistically significant improvement by carbidopa-levodopa treatment in any of: dark adaptation; BCVA; LLVA; drusen or reticular pseudodrusen measured by spectral domain(SD) optical coherence tomography(OCT)

Measurements:

1. Demographics at Visit 1;
2. Medical History and Physical Examination at Visit 1;
3. Electrocardiogram(ECG), complete blood count(CBC), Chem 20 and HbA1C at Visit 1;
4. Vital signs at Visits 1,3,4,5 and 6;
5. Non-directed assessment of adverse events at Visits 1,2, 3 and 4;
6. Ophthalmic history and comprehensive eye examination, including dark adaptation and SD OCT at Visit 2 (Baseline);
7. Low luminance questionnaire at visits 2, 3 and 4;
8. Pill count at Visits 3 and 4;
9. Re-measurement of dark adaptation, visual acuity under normal and low light conditions and SD OCT at Visits 3 and 4 (End of Study);

Statistics: Analysis of Variance with Independent Variables:

1. Active Drug vs Placebo;
2. Logarithm of daily dose of active drug;
3. Duration of treatment (measurements at Visits 3, 4, 5 and 6.

ELIGIBILITY:
1. Inclusion Criteria:

   * - A diagnosis of intermediate or advanced dry AMD in at least one eye. The other eye may be normal or have any stage of AMD.
   * - If the participant is taking AREDS vitamin supplements, these supplements must be continued for the duration of the study. If the participant is not taking AREDS vitamin supplements, these supplements must not be started during the study.
2. Exclusion Criteria:

   * - Any previous prescription for L-DOPA or dopamine agonist medications, or any planned use of any of these agents, except for study medication, during the study;
   * - Concurrent use of monoamine oxidase (MAO) inhibitors;
   * - With the exception of AMD or cataract or previous cataract operation; any eye condition, disease, history of surgery, or trauma in either eye, which can impair vision;
   * - Neurologic conditions which can impair vision;
   * - Parkinson's Disease;
   * - Dark adaptation rod intercept < 6.5 minutes;
   * - Significant orthostatic hypotension, defined as a drop in systolic blood pressure, immediately upon changing from the supine to standing position, of >19 mmHg, or a symptomatic drop in systolic blood pressure, immediately upon changing from the supine to standing position;
   * - Significant ECG abnormalities, as judged by the Investigator;
   * - Estimated glomerular filtration rate (eGFR) <30 ml/min;
   * - Liver enzymes >3 X the upper limit of normal;
   * - HbA1C >9.0;
   * - Any other significant lab abnormalities, as judged by the Investigator.
   * - Women with childbearing potential;
   * -Subjects who are not fluent in English.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | 90 +- 10 days
  Treatment Emergent Adverse Events (AEs) will be assessed at each visit. These will be classified as mild, moderate or severe and by body organ system. All AEs will be specifically reassessed at each subsequent visit. Serious AEs will be reported to the institutional Review Board(IRB). All AEs will be aggregated by treatment arm.

SECONDARY OUTCOMES:
Change from Baseline in Best Corrected Visual Acuity | 45 +/- 5 days and 90 +/- 10 days
  After refraction to ascertain that the participant has the optimum correction for refractive error, standard visual acuity testing will be performed with an ETDRS chart. Results will be ascertained at 45 +/-5 and 90 +/- 10 days, due to different dosing during the first and second 45 day periods. Results will be aggregated by treatment arm and treatment period.
Change from Baseline in Low Light Visual Acuity | 45 +/- 5 days and 90 +/- 10 days
  Using lenses for optimum correction for refractive error, Standard visual acuity testing will be performed using an ETDRS chart under standardized low light conditions. Results will be ascertained at 45 +/- 5 and 90 +/- 10 days, due to different dosing during the first and second 45 day periods. Results will be aggregated by treatment arm and treatment period.
Change from Baseline in Dark Adaptation | 45 +/- 5 days and 90 +/- 10 days
  Using an AdaptDX machine, using standardized intensity and duration of bright light, measurement of the time after bright light exposure required to adapt to dim light will be measured using rod intercept as the measurement. Results will be ascertained at 45 +/- 5 and 90 +/- 10 days, due to different dosing during the first and second 45 day periods. Results will be aggregated by treatment arm and treatment period.
Change from Baseline in Low Luminance Questionnaire Scores | 45 +/- 5 days and 90 +/- 10 days
  This will be measured using a standard questionaire evaluating ability to function in low light conditions. Results will be tabulated by all correct answers and by number of correct answers on each subscale. Results will be ascertained at 45 +/- 5 and 90 +/- 10 days, due to different dosing during the first and second 45 day periods. Results will be aggregated by treatment arm and treatment period.
Change from Baseline in Optical Coherence Tomography | 45 +/- 5 days and 90 +/- 10 days
  Evaluating retinal structure, including drusen and reticular pseudodrusen using a standard scanning laser device. Results will be ascertained at 45 +/- 5 and 90 +/- 10 days, due to different dosing during the first and second 45 day periods. Results will be aggregated by treatment arm and treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Snyder, MD, PhD, Principal Investigator — Robert W Snyder, MD, PhD, PC; Timothy C Fagan, MD, Study Director — Robert W Snyder, MD, PhD, PC
Locations (1):
- Robert W Snyder, MD, PhD, PC, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Jager RD, Mieler WF, Miller JW. Age-related macular degeneration. N Engl J Med. 2008 Jun 12;358(24):2606-17. doi: 10.1056/NEJMra0801537. No abstract available. PMID 18550876
- [Background] Bressler SB, Munoz B, Solomon SD, West SK; Salisbury Eye Evaluation (SEE) Study Team. Racial differences in the prevalence of age-related macular degeneration: the Salisbury Eye Evaluation (SEE) Project. Arch Ophthalmol. 2008 Feb;126(2):241-5. doi: 10.1001/archophthalmol.2007.53. PMID 18268216
- [Background] Nowacka B, Lubinski W, Honczarenko K, Potemkowski A, Safranow K. Ophthalmological features of Parkinson disease. Med Sci Monit. 2014 Nov 11;20:2243-9. doi: 10.12659/MSM.890861. PMID 25387009
- [Background] Ferrara N. Vascular endothelial growth factor and age-related macular degeneration: from basic science to therapy. Nat Med. 2010 Oct;16(10):1107-11. doi: 10.1038/nm1010-1107. No abstract available. PMID 20930754
- [Background] Kauppinen A, Paterno JJ, Blasiak J, Salminen A, Kaarniranta K. Inflammation and its role in age-related macular degeneration. Cell Mol Life Sci. 2016 May;73(9):1765-86. doi: 10.1007/s00018-016-2147-8. Epub 2016 Feb 6. PMID 26852158
- [Background] Lopez VM, Decatur CL, Stamer WD, Lynch RM, McKay BS. L-DOPA is an endogenous ligand for OA1. PLoS Biol. 2008 Sep 30;6(9):e236. doi: 10.1371/journal.pbio.0060236. PMID 18828673
- [Background] Falk T, Congrove NR, Zhang S, McCourt AD, Sherman SJ, McKay BS. PEDF and VEGF-A output from human retinal pigment epithelial cells grown on novel microcarriers. J Biomed Biotechnol. 2012;2012:278932. doi: 10.1155/2012/278932. Epub 2012 Apr 2. PMID 22547925
- [Background] Brilliant MH, Vaziri K, Connor TB Jr, Schwartz SG, Carroll JJ, McCarty CA, Schrodi SJ, Hebbring SJ, Kishor KS, Flynn HW Jr, Moshfeghi AA, Moshfeghi DM, Fini ME, McKay BS. Mining Retrospective Data for Virtual Prospective Drug Repurposing: L-DOPA and Age-related Macular Degeneration. Am J Med. 2016 Mar;129(3):292-8. doi: 10.1016/j.amjmed.2015.10.015. Epub 2015 Oct 30. PMID 26524704
- [Background] Sinemet package insert (FDA approved).
- [Background] Chandramohan A, Stinnett SS, Petrowski JT, Schuman SG, Toth CA, Cousins SW, Lad EM. VISUAL FUNCTION MEASURES IN EARLY AND INTERMEDIATE AGE-RELATED MACULAR DEGENERATION. Retina. 2016 May;36(5):1021-31. doi: 10.1097/IAE.0000000000001002. PMID 26925551
- [Background] Owsley C, McGwin G Jr, Clark ME, Jackson GR, Callahan MA, Kline LB, Witherspoon CD, Curcio CA. Delayed Rod-Mediated Dark Adaptation Is a Functional Biomarker for Incident Early Age-Related Macular Degeneration. Ophthalmology. 2016 Feb;123(2):344-351. doi: 10.1016/j.ophtha.2015.09.041. Epub 2015 Oct 30. PMID 26522707
- [Background] Wu Z, Ayton LN, Luu CD, Guymer RH. Longitudinal changes in microperimetry and low luminance visual acuity in age-related macular degeneration. JAMA Ophthalmol. 2015 Apr;133(4):442-8. doi: 10.1001/jamaophthalmol.2014.5963. PMID 25632841
- [Background] Hongyang Zhang; Nizar Saleh Abdelfattah; David S Boyer; Srinivas R Sadda, Longitudinal Quantitative OCT Analysis of Drusen in the Fellow Eye of Patients with Unilateral Neovascular Age-Related Macular Degeneration, ARVO Annual Meeting Abstract, 2015.
- [Background] Finger RP, Chong E, McGuinness MB, Robman LD, Aung KZ, Giles G, Baird PN, Guymer RH. Reticular Pseudodrusen and Their Association with Age-Related Macular Degeneration: The Melbourne Collaborative Cohort Study. Ophthalmology. 2016 Mar;123(3):599-608. doi: 10.1016/j.ophtha.2015.10.029. Epub 2015 Dec 8. PMID 26681391
- [Background] Owsley C, McGwin G, Jackson GR, Heimburger DC, Piyathilake CJ, Klein R, White MF, Kallies K. Effect of short-term, high-dose retinol on dark adaptation in aging and early age-related maculopathy. Invest Ophthalmol Vis Sci. 2006 Apr;47(4):1310-8. doi: 10.1167/iovs.05-1292. PMID 16565362
- [Background] Westfall, T.C. and Westfall, D.P. Drugs Acting at Synaptic and Neuroeffector Junctions. Pharmacological Basis of Therapeutics, 11th Edition, 530-535, McGraw-Hill, 2006.
- [Background] Standaert, D.G. and Young, A.B. Treatment of Central Nervous System Degenerative Disorders. Pharmacological Basis of Therapeutics, 11th Edition, 530-535, McGraw-Hill, 2006.